CLINICAL TRIAL: NCT00583869
Title: The Role of Pregabalin in the Treatment of Post-Operative Pain in Fracture Patients
Brief Title: Role of Pregabalin in Treatment of Post-Op Pain in Fracture Patients
Acronym: LYRICA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F061204006
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2012-05

CONDITIONS: Post-operative Pain
Keywords: Post-operative Pain; Fracture Patients; Pregabalin; LYRICA
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Patient to receive placebo beginning on the day of surgery until discharge.
  Interventions: Drug: Placebo
- 2 (Experimental): Patient to receive 75mg PO BID pregabalin beginning on the day of surgery until discharge.
  Interventions: Drug: Pregabalin
- 3 (Experimental): Patient to receive 150mg PO BID pregabalin beginning on the day of surgery until discharge.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Placebo — Two hours before surgery, patients will receive 75mg of pregabalin. Patients will be placed on a patient-controlled anesthesia pump (PCA) for 24 hours. On post-operative day one, the patients will be switched to oral oxycodone as needed with supplementation with IV Demerol for breakthrough pain. In addition, patients will receive a placebo PO BID beginning on the day of surgery until discharge.
  Upon discharge, the patient will be given study medication (placebo PO BID). Rescue medications will be allowed during the study (including post-operative and outpatient periods). Outpatient rescue medications will consist of hydrocodone/APAP 7.5mg PO Q6H PRN. Patients will be followed for three months as an outpatient.
  Arms: 1
Drug: Pregabalin — Two hours before surgery, patients will receive 75mg of pregabalin. Patients will be placed on a patient-controlled anesthesia pump (PCA) for 24 hours. On post-operative day one, the patients will be switched to oral oxycodone as needed with supplementation with IV Demerol for breakthrough pain. In addition, patients will receive 75mg PO BID beginning on the day of surgery until discharge.
  Upon discharge, the patient will be given study medication (pregabalin 75mg PO BID). Rescue medications will be allowed during the study (including post-operative and outpatient periods). Outpatient rescue medications will consist of hydrocodone/APAP 7.5mg PO Q6H PRN. Patients will be followed for three months as an outpatient.
  Other Names: LYRICA
  Arms: 2
Drug: Pregabalin — Two hours before surgery, patients will receive 75mg of pregabalin. Patients will be placed on a patient-controlled anesthesia pump (PCA) for 24 hours. On post-operative day one, the patients will be switched to oral oxycodone as needed with supplementation with IV Demerol for breakthrough pain. In addition, patients will receive 150mg PO BID beginning on the day of surgery until discharge.
  Upon discharge, the patient will be given study medication (pregabalin 150mg PO BID). Rescue medications will be allowed during the study (including post-operative and outpatient periods). Outpatient rescue medications will consist of hydrocodone/APAP 7.5mg PO Q6H PRN. Patients will be followed for three months as an outpatient.
  Other Names: LYRICA
  Arms: 3

SUMMARY:
This is a randomized, prospective, double-blind pilot study designed to evaluate the potential effectiveness of pregabalin in post-operative pain management for patients who have sustained a fracture.

DETAILED DESCRIPTION:
On admission, all patients who have sustained orthopaedic injuries of any type, including pelvis, will be screened. However, only those patients who will undergo a single episode of surgery during this hospitalization to surgically repair only one of their orthopaedic fractures will be interviewed by a clinical research nurse. If the patient meets all criteria for inclusion/exclusion in the study, the attending physician will consent the patient for inclusion in the study. Upon enrollment into the study, the clinical research nurse will obtain a thorough history from the patient concerning prior narcotic use, response to painful events in the past and will record details of the injury. Prior to surgery, the patient will be treated with narcotic pain medication as required in the judgment of the attending physician. The patient will then be randomized before surgery into a placebo group or pregabalin group. The attending physician will be blinded as to which study arm the patient is in.

Two hours before surgery, patients will receive 75mg of pregabalin. Patients will be placed on a patient-controlled anesthesia pump (PCA) for 24 hours. On post-operative day one, the patients will be switched to oral oxycodone as needed with supplementation with IV Demerol for breakthrough pain. In addition, patients will receive either pregabalin 75mg orally (PO) BID, pregabalin 150mg PO BID or placebo beginning on the day of surgery until discharge.

The clinical research nurse will complete a form which records the daily use of each of the post-operative pain medications. She will also ask the patient to complete a Visual Analog Scale (VAS) to assess pain each day while in the hospital.

Upon discharge, the patient will be given study medication (pregabalin, 75mg PO BID, 150mg PO BID or placebo). Rescue medications will be allowed during the study (including post-operative and outpatient periods). Outpatient rescue medications will consist of hydrocodone/acetamenophen (APAP) 7.5mg PO every sic hours (Q6H) as needed (PRN). Patients will be followed for three months as an outpatient.

ELIGIBILITY:
Inclusion Criteria:

* fractures requiring operative treatment during a single operative episode
* Adult patients between the ages of 19 and 70

Exclusion Criteria:

* prior medical history of narcotic abuse or narcotic use within 2 weeks of injury (except those given in hospital)
* contraindications to pregabalin or narcotic analgesics
* significant closed head injury
* psychiatric illness requiring medical treatment
* surgery for other injuries (splenectomy, etc)
* history of seizures requiring current anticonvulsant therapy
* inability or unwillingness to give informed consent

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Amount of pain medication in morphine equivalent units used during the hospitalization. | Screening - 5 - 15 minutes; Consent - 5-15 minutes; Follow-up - three 15-30-minute visits

SECONDARY OUTCOMES:
Secondary outcome measures will include Visual Analog Score, timing and frequency of rescue medications, Short-Form 36 Health Survey scores, and adverse events. | Three 15-30-minute visits after surgery to complete SF-36 and Visual Analog Score for Pain.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Theiss, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Turan A, White PF, Karamanlioglu B, Memis D, Tasdogan M, Pamukcu Z, Yavuz E. Gabapentin: an alternative to the cyclooxygenase-2 inhibitors for perioperative pain management. Anesth Analg. 2006 Jan;102(1):175-81. doi: 10.1213/01.ane.0000184824.43411.63. PMID 16368826
- [Background] Fischer HB, Simanski CJ. A procedure-specific systematic review and consensus recommendations for analgesia after total hip replacement. Anaesthesia. 2005 Dec;60(12):1189-202. doi: 10.1111/j.1365-2044.2005.04382.x. PMID 16288617
- [Background] Sills GJ. The mechanisms of action of gabapentin and pregabalin. Curr Opin Pharmacol. 2006 Feb;6(1):108-13. doi: 10.1016/j.coph.2005.11.003. Epub 2005 Dec 22. PMID 16376147